CLINICAL TRIAL: NCT05062265
Title: Internal Brace Augmented Anterior Inferior Tibiofibular Ligament Repair and Its Post-operative Effects on Syndesmotic Volumes: A Prospective, Single-blinded, Randomized Study
Brief Title: Internal Brace Augmented Anterior Inferior Tibiofibular Ligament Repair: Post-operative Syndesmotic Volumes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vann Virginia Center for Orthopaedics dba Atlantic Orthopaedic Specialists (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Blake E. Moore, MD, Principal Investigator, Vann Virginia Center for Orthopaedics dba Atlantic Orthopaedic Specialists
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: AOS-0001
Record Dates: First submitted 2021-07-27; First posted 2021-09-30 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Syndesmotic Injuries; Ligament Rupture; Bimalleolar Fractures; Trimalleolar Fractures
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tight Rope Fixation (Active Comparator)
  Interventions: Device: Tight rope fixation
- tight rope fixation w/ AITFL repair augmentation with an internal brace (Active Comparator)
  Interventions: Device: Tight rope fixation with an anterior inferior tibiofibular ligament (AITFL) repair augmentation with an internal brace

INTERVENTIONS:
Device: Tight rope fixation — a traditional tight rope fixation is performed on one randomized set of subjects
  Arms: Tight Rope Fixation
Device: Tight rope fixation with an anterior inferior tibiofibular ligament (AITFL) repair augmentation with an internal brace — A tight rope fixation with an anterior inferior tibiofibular ligament (AITFL) repair augmentation with an internal brace set of subjects to compare syndesmotic volume
  Arms: tight rope fixation w/ AITFL repair augmentation with an internal brace

SUMMARY:
Over the course of a year from the start of the research study, twenty subjects will be randomized evenly into one of two groups after an informed consent is obtained: a traditional tight rope fixation group or a tight rope fixation with an anterior inferior tibiofibular ligament (AITFL) repair augmentation with an internal brace group. Postoperative reduction was assessed by 3D volumetric ratios and measured by weight-bearing CT at 6-weeks and 3-months post-operation. Patient Reported Outcomes (PROs) were collected preoperatively, and at 6-weeks, 3-months, 6-months, and 1-year post-operation and included the Foot and Ankle Outcome Score and the 36-Item Short Form Survey Instrument (RAND-36) . Differences in volumetric ratios and PROs were evaluated between groups and time periods.

ELIGIBILITY:
Inclusion Criteria:

* patients who fit the study injury list

Exclusion Criteria:

* smokers
* prior surgery on ankle
* bi-lateral surgery
* recent participation in another study within the last 90days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blake E Moore, MD, Principal Investigator — Vann Virginia Center for Orthopaedics dba Atlantic Orthopaedic Specialists; Ashley Suttmiller, PhD, Study Chair — Clinical Researcher; Brice A Snyder, MSAT, Study Director — Director of Clinical Research
Locations (1):
- Atlantic Orthopaedic Specialists, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n = 2)
  - Not meeting inclusion criteria: Intact AITFL (n = 2)
Groups:
- Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace: Tight rope fixation with an anterior inferior tibiofibular ligament (AITFL) repair augmentation with an internal brace: A tight rope fixation with an anterior inferior tibiofibular ligament (AITFL) repair augmentation with an internal brace
Period: Overall Study
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Started | 12 | 9
Completed | 11 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (13.3) | 55.9 (19.3) | 52.9 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20
Height (m) [Mean (Standard Deviation); unit: meters] | 1.6 (0.1) | 1.7 (0.1) | 1.7 (0.5)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 85.0 (16.0) | 81.0 (13.0) | 83.3 (14.5)
Operative Side [Count of Participants; unit: Participants]
  Left | 5 | 3 | 8
  Right | 6 | 6 | 12
FAOS- Pain [Mean (Standard Deviation); unit: units on a scale] | 20.2 (19.2) | 30.7 (20.9) | 25 (20.3)
FAOS- Symptoms [Mean (Standard Deviation); unit: units on a scale] | 26.9 (21.9) | 40.8 (23.4) | 33 (23)
FAOS- Daily Life [Mean (Standard Deviation); unit: units on a scale] | 19 (19) | 33 (22) | 25 (21)
FAOS- Sports/Rec [Mean (Standard Deviation); unit: units on a scale] | 7.3 (12.5) | 6.1 (9.9) | 7 (11.2)
FAOS- QoL [Mean (Standard Deviation); unit: units on a scale] | 6 (14) | 10 (13.6) | 8 (13.6)
RAND-36 PHC [Mean (Standard Deviation); unit: units on a scale] — 36-Item Short Form Survey Instrument (RAND-36 or SF-36) Physical Health Component (PHC)
  units on a scale | 37.2 (11.2) | 39.1 (10.7) | 38.1 (11)
RAND-36 MHC [Mean (Standard Deviation); unit: units on a scale] — 36-Item Short Form Survey Instrument (SF-36 or RAND-36) Mental Health Component (MHC)
  units on a scale | 46.8 (11.2) | 51.0 (7.7) | 48.7 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Syndesmotic Volumetric Ratio
Description: use of weight-bearing CT scan to measure; In order to compare the 3D syndesmotic volume between groups, the volume ratio was calculated for each patient by dividing the syndesmotic volume of the operative ankle by the syndesmotic volume of the contralateral uninjured ankle
Time Frame: 6-Weeks Post-op
Measure: Mean (Standard Deviation); unit: Volumetric Ratio
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
Volumetric Ratio | 1.2 (0.2) | 1.1 (0.1)

2. Primary Outcome: Syndesmotic Volumetric Ratio
Description: as for outcome 1
Time Frame: 3 months post-operative volume
Measure: Mean (Standard Deviation); unit: Volumetric Ratio
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
Volumetric Ratio | 1.2 (0.3) | 1.1 (0.3)

3. Secondary Outcome: 36-Item Short Form Survey Instrument (RAND-36) Summary Scores
Description: The RAND-36 is a health-related quality-of-life questionnaire consisting of 36 questions that measure eight health domains to assess physical and mental health. Scores are 00-100. Higher scores equate to better quality of life and inverse for lower scores. The Physical Health Component and Mental Health Component summary scores were calculated using the oblique method to reduce the risk of underrepresenting mental health scores.
Time Frame: 6 weeks post-operative
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
score on a scale
  PHC | 35.2 [30 to 45] | 36.3 [32 to 41]
  MHC | 45.3 [39 to 52] | 47.6 [43 to 52]

4. Secondary Outcome: RAND-36 Summary Scores
Description: The Short Form-36 (SF-36 or RAND-36) is a health-related quality-of-life questionnaire consisting of 36 questions that measure eight health domains to assess physical and mental health. Scores are 00-100. Higher scores equate to better quality of life and inverse for lower scores. The Physical Health Component and Mental Health Component summary scores were calculated using the oblique method to reduce the risk of underrepresenting mental health scores.
Time Frame: 3 months post-operative
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
score on a scale
  PHC | 50.7 [44 to 58] | 44.5 [37 to 52]
  MHC | 52.2 [46 to 59] | 52.8 [47 to 58]

5. Secondary Outcome: RAND-36 Summary Scores
Description: The SF-36 is a health-related quality-of-life questionnaire consisting of 36 questions that measure eight health domains to assess physical and mental health. Scores are 00-100. Higher scores equate to better quality of life and inverse for lower scores. The Physical Health Component and Mental Health Component summary scores were calculated using the oblique method to reduce the risk of underrepresenting mental health scores.
Time Frame: 6 months post-operative
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
score on a scale
  PHC | 48.5 [42 to 55] | 51.9 [45 to 59]
  MHC | 51.3 [45 to 57] | 55.8 [53 to 59]

6. Secondary Outcome: RAND-36 Summary Scores
Description: as for outcome 5
Time Frame: 1 year post-operative
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
score on a scale
  PHC | 49.7 [44 to 55] | 51 [43 to 59]
  MHC | 53.3 [48 to 59] | 54.9 [50 to 60]

7. Secondary Outcome: Foot and Ankle Outcome Score (FAOS)
Description: FAOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport(Rec), and foot and ankle-related Quality of Life (QOL). The last week is taken into consideration when answering the questionnaire. Standardized answer options are given (% Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: 6 weeks post-operative
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
units on a scale
  Pain | 53.1 [35 to 71] | 71.6 [55 to 88]
  Symptoms | 56.4 [44 to 69] | 69.6 [58 to 82]
  Daily Life | 60.5 [45 to 76] | 72.6 [58 to 87]
  Sports/Rec | 17.3 [0 to 38] | 42.8 [14 to 71]
  QoL | 29.5 [15 to 45] | 38.3 [12 to 65]

8. Secondary Outcome: Foot and Ankle Outcome Score (FAOS)
Description: as for outcome 7
Time Frame: 3 months post-operative
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
units on a scale
  Pain | 70.7 [57 to 84] | 74.8 [57 to 93]
  Symptoms | 69.1 [60 to 79] | 69.6 [58 to 81]
  Daily Life | 80 [69 to 91] | 78 [63 to 93]
  Sports/Rec | 46.8 [24 to 69] | 55.6 [30 to 82]
  QoL | 46.3 [30 to 63] | 41.2 [25 to 58]

9. Secondary Outcome: Foot and Ankle Outcome Score (FAOS)
Description: as for outcome 7
Time Frame: 6 months post-operative
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
units on a scale
  Pain | 70 [55 to 85] | 82.8 [70 to 95]
  Symptoms | 62 [50 to 74] | 80.1 [72 to 88]
  Daily Life | 75.1 [59 to 91] | 89.3 [79 to 100]
  Sports/Rec | 45 [22 to 68] | 72.8 [55 to 91]
  QoL | 46.8 [29 to 65] | 64 [53 to 75]

10. Secondary Outcome: Foot and Ankle Outcome Score (FAOS)
Description: as for outcome 7
Time Frame: 1 year post-operative
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
Number analyzed (Participants) | 11 | 9
units on a scale
  Pain | 80.5 [70 to 91] | 87 [75 to 99]
  Symptoms | 73.6 [62 to 85] | 80.3 [67 to 94]
  Daily Life | 87.1 [78 to 96] | 90.8 [81 to 100]
  Sports/Rec | 63.2 [43 to 84] | 77.2 [58 to 97]
  QoL | 63.2 [49 to 77] | 73.8 [58 to 89]

ADVERSE EVENTS:
Time Frame: 1 year follow up from surgery date.
Arm/Group | Tight Rope Fixation | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tight Rope Fixation (N=12) | Tight Rope Fixation w/ AITFL Repair Augmentation With an Internal Brace (N=9)
Post-operative Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Post-operatively, subject had persistent lateral lower leg pain and determined to have painful hardware. Subject's hardware from the indexed surgery was removed during the study follow up phase via second surgery and had resolution of pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT05062265/Prot_SAP_000.pdf